CLINICAL TRIAL: NCT00219505
Title: Effect of Acupuncture on Symptoms of Diarrhea and Pain in Diarrhea Predominant Irritable Bowel Syndrome (IBS) and Effect on Plasma Beta-endorphin and Serotonin Levels.
Brief Title: Effect of Acupuncture on Symptoms of Diarrhea and Pain in IBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible subjects identified during recruitment
Sponsor: Penn State University (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2000-343
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diarrhea-predominant irritable bowel syndrome; Acupuncture; abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: acupuncture

SUMMARY:
Acupuncture has been used for centuries in China in the treatment of diarrhea. Our hypothesis is that acupuncture is effective in the treatment of abdominal pain and diarrhea in patients with diarrhea-predominant IBS

DETAILED DESCRIPTION:
Patients will complete a diary to determine if they qualify for the study. Patients will be randomized to receive either acupuncture or sham acupuncture (needle insertion 1 cm away from acupuncture site). Patients will be blinded to whether they are receiving acupuncture or sham acupuncture. The acupuncturist is blinded as to the patient response. The patients will undergo venupuncture to draw blood to determine sertotonin and beta-endorphin levels. They will receive treatment in 12 sessions over 4 weeks. They will maintain a diary during this time period to document level of pain and frequency of bowel movements. Blood will be drawn at week 2 and 4 and, 6 weeks after cessation of treatment, subjects will again record abdominal symptoms and frequency of bowel movements for 2 weeks. Blood will be drawn for hormone levels at 8 weeks after completion of study.

ELIGIBILITY:
Inclusion Criteria:

* frequence of bowel movement of at least 3/day
* global disease severity of at least 3

Exclusion Criteria:

* taking medications which will influence frequency of bowel movement
* patient taking anticoagulants or suffering from coagulopathy
* pregancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2001-08; Study Completion 2004-01

PRIMARY OUTCOMES:
Frequency of bowel movement

SECONDARY OUTCOMES:
Abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ouyangm, MD, Principal Investigator — Penn State College of Medicine and Penn State Milton S. Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States